CLINICAL TRIAL: NCT07270029
Title: Sensory Toys for Anxiety Reduction - Can Fidget Toys Improve Stress and Help Children to Cope Before Surgery (STARFISH)
Acronym: STARFISH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Telethon Kids Institute (Other)
Collaborators: Child and Adolescent Health Service - Perth (Other Government); University of Sao Paulo (Other); Hospital das Clínicas de São Paulo - SP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RGS0000007990
Record Dates: First submitted 2025-11-13; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Perioperative Anxiety
Keywords: children; pediatrics; surgery; pediatric anaesthesia; anxiety; perioperative anxiety; fidget toys; sensory toys
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised controlled multicentre trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory toy group (Experimental): Children receive a sensory toy of their choice preoperatively
  Interventions: Other: Pre-operative sensory toy
- Control group (Sham Comparator): Children receive a sensory toy at the time of discharge from hospital
  Interventions: Other: Post-operative sensory toy

INTERVENTIONS:
Other: Pre-operative sensory toy — Sensory toy (e.g., spinners, putty, stability balls) chosen by the child on the day of surgery pre-operatively. All sensory toys will be sourced from Australian company for Perth Children's Hospital and from a Brazilian company for Hospital das Clinicas HCFMUSP.
  Other Names: Fidget toy; fidget device
  Arms: Sensory toy group
Other: Post-operative sensory toy — Sensory toy (e.g., spinners, putty, stability balls) chosen by the child upon discharge from hospital following their surgery. All sensory toys will be sourced from Australian company for Perth Children's Hospital and from a Brazilian company for Hospital das Clinicas HCFMUSP.
  Other Names: fidget toy; fidget device
  Arms: Control group

SUMMARY:
Anxiety associated with medical procedures is common, with 40-80% of children experiencing significant symptoms and postoperative consequences, including distress and delirium, increased intensity/duration of pain, prolonged hospital stays, behavioural/sleep disturbance and avoidance of medical encounters, which often remain into adulthood.

Extensive consumer research has shown that a key priority for Australian consumers of all ages in relation to paediatric hospital care is addressing the fear and anxiety in children throughout the hospital experience (second only to anaesthesia safety for adults and third following anaesthesia safety and pain management for children).

The STARFISH trial was driven by our consumer partners, particularly our youth consumers. It is well known that distraction is a coping strategy that can help with perioperative anxiety, and all members of the perioperative team commonly employ distraction techniques with patients during routine clinical care. One potential form of distraction involves sensory activities - fidget devices or sensory toys such as spinners, putty, and stability balls are increasingly being used within school settings to help students academically and behaviourally, with applicability for neurodiverse (e.g., autistic, Attention Deficit Hyperactivity Disorder (ADHD)) children being one area of particular interest. However, the research behind sensory toys is inconclusive.

Sensory toys have been suggested to our team-from numerous consumers of all ages, including neurodiverse and neurotypical consumers-as a method to reduce anxiety in the preoperative period, thus leading to the design of the STARFISH trial.

This project aims to assess the use of a sensory toy (of the child's choice) in the perioperative period on the day of surgery to reduce perioperative anxiety and distress.

DETAILED DESCRIPTION:
Anxiety associated with hospital experiences is common and a key concern for families and clinicians. Anxiety is linked to a number of adverse outcomes in children, including an increased risk of emergence delirium after anaesthesia, increased/prolonged pain, increased medication use (particularly strong pain killers, sedating agents), prolonged hospital stay, negative post-procedural behavioural outcomes, distress to children, families and medical staff, as well as distress to other children and families who witness a child in distress. Furthermore, anxiety can lead to long-term avoidance of healthcare encounters and consequently to negative health outcomes which can be life-long. This avoidance can impact not only the child's health care trajectory but also the health-trajectory and wellbeing of their parents and siblings.

In many institutions, including Perth Children's Hospital (PCH), pharmacological interventions in the form of sedative pre-medication are currently the most common strategy used to manage preoperative anxiety. Midazolam, for example, is a pre-medication widely used to reduce preoperative anxiety. Various studies have displayed the efficacy of midazolam in improving child behaviour during induction and reducing anxiety. Pharmacological interventions, however, have limitations, including the requirement to monitor patients after drug administration for potential adverse side effects and changes in vital signs. This increases staff requirements, placing more pressure on nurses and driving costs upwards. Paediatric patients may even find the process of taking pre-medication more traumatising than the hospital experience itself. Furthermore, while children may seem less anxious during the induction of anaesthesia following premedication with midazolam, research suggests that midazolam can paradoxically increase the incidence of post-hospital behavioural change. Some patients describe feeling anxious inside and "locked in", while from the outside looking calm, increasing their perceived anxiety even more. Additionally, pre-medication does not address the cause of the anxiety or help to develop strategies that may improve a child's ability to cope with stressful circumstances into the future.

A promising strategy that can reduce intense anxiety is distraction, and it has long been recognised that distraction leads to a significant reduction in perioperative anxiety. Distraction can take many forms, and while it is an under-researched area, there is a high potential for involving distraction via sensory experiences.

In this context, the use of sensory toys (e.g., spinners, putty, and stability balls) has been repeatedly suggested by consumers of all ages to aid with anxiety management. The benefit of sensory toys is that they can be used by nearly all children of a certain age group, including many who are neurodiverse, have special needs, and children from diverse cultural backgrounds, languages other than English, and those in regional/remote areas. Previous attempts at delivering tools for children to self-manage symptoms of anxiety have been labour-intensive to implement and train. Although purchasing the sensory toy incurs a cost, it remains a relatively inexpensive intervention that, could be easily implemented to benefit the child beyond the hospital experience. The costs are likely offset by a reduced requirement for premedication and thus a lower requirement for close nursing observation levels and time savings due to fewer theatre delays caused by incorrect timing of premedications.

This randomised controlled multicentre trial will assess the effect of a sensory toy on the child's preoperative anxiety, administered on the day of surgery. It will further assess, the cost of the intervention, the impact on anaesthesia induction, premedication as well as immediate and short term (1 week) outcomes for children undergoing surgery or procedures under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-15.99 years of age
* Children admitted to the day of surgery unit undergoing elective surgery at Perth Children's Hospital or Hospital das Clinicas HCFMUSP as day case surgeries or with a maximum hospital stay of one night postoperatively

Exclusion Criteria:

* Children coming for surgery via wards other than the day of surgery unit
* Language barriers impeding data collection
* Department for Child Protection and Family Support is involved in the care of the child
* Inability for the child to interact with the sensory toy safely, such as children with severe global developmental delay (GDD).

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Compare anxiety levels on day of surgery at sign-in to theatre (T2, when patient is moved from pre-operative ward to induction room) and baseline (T1, on pre-operative ward ) between children in sensory toy group and those in the control group. | Baseline anxiety will be assessed on the preoperative ward on the day of surgery (on pre-operative ward, T1), and at sign-in to theatre (when patient is moved from pre-operative ward to induction room, T2 ).
  Anxiety will be measured using the modified Yale Perioperative Anxiety Scale (mYPAS). mYPAS consists of 22 items in 5 categories: activity (4 items), vocalisations (6 items), emotional expressivity (4 items), state of apparent arousal (4 items) and use of parents (4 items). The highest observed behavioural item in each category is the score for that category. The minimum score at each timepoint is 5 and the maximum score is 22. High mYPAS scores at each time point are indicative of higher preoperative anxiety.

SECONDARY OUTCOMES:
Compare anxiety levels at baseline, sign in to theatre, and at induction of anaesthesia on the day of surgery between the sensory toy group and control group | Anxiety will be assessed on the day of surgery in the perioperative holding area (T1, in pre-operative holding area), at sign-in to theatre (T2,when patient is moved from ward to induction room) and during induction (T3, when mask or needle is applied)
  Anxiety will be measured using the modified Yale Perioperative Anxiety Scale (mYPAS). mYPAS consists of 22 items in 5 categories: activity (4 items), vocalisations (6 items), emotional expressivity (4 items), state of apparent arousal (4 items) and use of parents (4 items). The highest observed behavioural item in each category is the score for that category. The minimum score at each timepoint is 5 and the maximum score is 22. High mYPAS scores at each time point are indicative of higher preoperative anxiety.
Compare induction compliance between the sensory toy group and the control group on the day of surgery | Assessed on the day of surgery during anaesthetic induction (application of the mask or the needle)
  Induction compliance will be assessed using the induction compliance checklist (ICC). The ICC contains 11 items, giving a score from 0 (extremely compliant) to 11 (extremely uncompliant).
Compare postoperative analgesia requirements between control group and sensory toy group | Analgesics will be recorded until 24 hours post-surgery or time of discharge, whichever is sooner.
  All post-operative analgesics (paracetamol, NSAIDs, opioids) given post-operatively will be recorded
Comparison of incidence of emergence delirium between sensory toy and control groups | Emergence delirium will be assessed after surgery when the child wakes immediately after anaesthesia until discharge from the post-anaesthetic care unit (PACU) on the day of surgery.
  Emergence delirium will be assessed by the post-operative recovery nurse using the WATCHA scale. The WATCHA scale is scored from 0 (asleep) to 4 (agitated, thrashing around) , scores greater than or equal to 3 on this scale are indicative of emergence delirium.
Compare post-operative behavioural outcomes between control group and sensory toy group | Assessed on days 1 and 7 post-operatively
  Assessed using the Post-Hospitalisation Behaviour Questionnaire for Ambulatory Surgery (PHBQ-AS). The PHBQ-AS consists of 11 questions regarding a patient's behaviour and is answered using a 5-point likert scale (much less than before, less than before, same as before, more than before, much more than before).
Assessment of the parental and child satisfaction with the intervention | Assessed on the day of surgery at sign-out to theatre (patient moved from ward to induction room) or prior to the administration of a sedative premedication; on the post-operative ward before hospital discharge, and at 7 days post-discharge
  Assessed on a 5-point Likert scale
Compare differences in anxiety, induction compliance, post-operative analgesia requirements, emergence delirium and post-operative behavioural outcomes between neurodiverse and neurotypical children | Neurodiversity will be assessed by a researcher via a questionnaire administered prior to surgery.
  Neurodiversity will be assessed via parent report of whether the child has a formal diagnosis of autism and/or ADHD, as well as parent completion of a brief item set based on DSM-5-TR criteria for autism and the Strength and Difficulties Questionnaire measure of ADHD in childhood as well as the Perth Autism Scale.
Compare incidence of emergence delirium between patients in the sensory toy group and control group | Emergence delirium will be assessed after surgery when the child wakes immediately after anaesthesia until discharge from the post-anaesthetic care unit (PACU) on the day of surgery.
  Emergence delirium will be assessed by the post-operative recovery nurse using the Pediatric Anaesthesia Emergence Delirium (PAED) scale in the post anaesthetic care unit (PACU). The PAED scale consists of 5 items and is scored on a 5 point scale (not at all, just a little, quite a bit, very much, extremely). higher scores are indicative of emergence delirium, the maximum score is 20 and minimum score is 0.
Compare incidence of perioperative respiratory adverse events (PRAE) and post-operative nausea and vomiting (PONV) between neurodiverse and neurotypical children | PRAE will be assessed by the anaesthetist during anaesthetic induction, maintenance and emergence and by the recovery nurse while in the post-anaesthetic care unit (PACU). PONV will be assessed from waking in PACU until 24 hours post-surgery or discharge
  Perioperative respiratory adverse events (PRAE) are defined as: Major PRAE: laryngospasm or bronchospasm (as determined by the anaesthetist or recovery nurse) or desaturation <85% SpO2 for more than 1 minute on pulse oximetry. Minor PRAE: desaturation (<95% SpO2 for more than 10 seconds on pulse oximetry), airway obstruction, severe coughing, post-operative stridor. Each individual PRAE (laryngospasm, bronchospasm, desaturation, airway obstruction, severe persistent coughing and post-operative stridor) will be considered separately. PONV will be assessed by observing any incidence of nausea or vomiting post-operatively, and any administration of antiemetic medication.
Compare the post-operative behavioural outcomes between patients in the sensory toy group and control group using the Paediatric Scale for Quality of Recovery (PedSQoR). | Assessed 1 day and 7 days post- surgery
  post-operative behavioural outcomes will be measured using the Paediatric Scale for Quality of Recovery (PedSQoR). The PedsQoR is made of 20 questions, the overall score ranges from 20 to 100 and higher scores indicate a better quality of recovery or more complete recovery.
Compare anxiety levels a baseline, sign in to theatre and at induction of anaesthesia on the day of surgery between neurodiverse and neurotypical children | Anxiety will be assessed on the day of surgery in the perioperative holding area (T1, in pre-opeative ward), at sign-in to theatre (T2, when patient is moved from ward to induction room) and during induction (T3, when mask or needle is applied).
  Anxiety will be measured using the modified Yale Perioperative Anxiety Scale. mYPAS consists of 22 items in 5 categories: activity (4 items), vocalisations (6 items), emotional expressivity (4 items), state of apparent arousal (4 items) and use of parents (4 items). The highest observed behavioural item in each category is the score for that category. The minimum score at each timepoint is 5 and the maximum score is 22. High mYPAS scores at each time point are indicative of higher preoperative anxiety.
Compare induction compliance on the day of surgery between neurodiverse and neurotypical children | Assessed on the day of surgery during anaesthetic induction
  Induction compliance will be assessed using the induction compliance checklist (ICC). The ICC contains 11 items, giving a score from 0 (extremely compliant) to 11 (extremely uncompliant).
Compare post-operative analgesia requirements between neurodiverse and neurotypical children | Analgesics will be recorded until 24 hours post-surgery or time of discharge from hospital
  All post-operative analgesics (paracetamol, NSAIDS, opioids) given post-operatively will be recorded.
Compare incidence of emergence delirium between neurodiverse and neurotypical children | Emergence delirium will be assessed after surgery when the child wakes immediately after anaesthesia until discharge from the post-anaesthetic care unit (PACU) on the day of surgery.
  Emergence delirium will be assessed by the post-operative recovery nurse using the WATCHA Scale. The WATCHA Scale is scored from 0 (asleep) to 4 (thrashing around). Scores greater than or equal to 2 on this scale are indicative of emergence delirium.
Compare incidence of emergence delirium between neurodiverse and neurotypical children | Emergence delirium will be assessed after surgery when the child wakes immediately after anaesthesia until discharge from the post-anaesthetic care unit (PACU) on the day of surgery.
  Emergence delirium will be assessed by the post-operative recovery nurse using the Pediatric Anaesthesia Emergence Delirium (PAED) scale in the post anaesthetic care unit (PACU). The PAED scale consists of 5 items and is scored on a 5 point scale (not at all, just a little, quite a bit, very much, extremely). higher scores are indicative of emergence delirium, the maximum score is 20 and minimum score is 0.
Compare post-operative behavioural outcomes between neurodiverse and neurotypical children | Assessed on days 1 and 7 post-operatively
  Assessed using the Post-Hospitalisation Behaviour Questionnaire for Ambulatory Surgery (PHBQ-AS). The PHBQ-AS consists of 11 questions regarding a patient's behaviour and is answered using a 5-point likert scale (much less than before, less than before, same as before, more than before, much more than before).
Compare the post-operative behavioural outcomes between neurodiverse and neurotypical children using the Paediatric Scale for Quality of Recovery (PedSQoR). | Assessed 1 day and 7 days post- surgery
  post-operative behavioural outcomes will be measured using the Paediatric Scale for Quality of Recovery (PedSQoR). The PedsQoR is made of 20 questions, the overall score ranges from 20 to 100 and higher scores indicate a better quality of recovery or more complete recovery.

CONTACTS AND LOCATIONS:
Locations (2):
- Perth Children's Hospital, Perth, Western Australia, Australia
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No